CLINICAL TRIAL: NCT07302594
Title: Effects of Oro-esophageal Versus Nasogastric Tubes on Swallowing Function in Ischemic Stroke Survivors: A Randomized Controlled Trial
Brief Title: Effects of Oro-esophageal Tubes on Swallowing Function in Ischemic Stroke Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Principle Investigator, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IOEvsNGonStroke
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oro-esophageal Feeding (Experimental): Patients will receive basic rehabilitation therapy in accordance with relevant guidelines. In addition, patients in this group will receive oro-esophageal tube feeding, with 3-6 feeding sessions per day. The feeding tube is inserted before each meal and removed immediately after feeding. Both groups of participants are administered the same nutritional standards.
  Interventions: Behavioral: standard rehabilitation therapy; Dietary Supplement: Oro-esophageal Feeding
- Nasogastric Feeding (Active Comparator): Patients will receive basic rehabilitation therapy in accordance with relevant guidelines. In addition, patients in this group will receive nasogastric tube feeding, with an interval of at least 2 hours between each feeding session. The feeding tube remains indwelling after insertion and is not removed. Both groups of participants are administered the same nutritional standards.
  Interventions: Behavioral: standard rehabilitation therapy; Dietary Supplement: Nasogastric Feeding

INTERVENTIONS:
Behavioral: standard rehabilitation therapy — Patients will receive corresponding interventions for secondary prevention in accordance with relevant guidelines and the conditions of each participating center, as well as common rehabilitation therapies. These interventions will be consistent between the two groups.
Dietary Supplement: Oro-esophageal Feeding — Before each feeding, inside and outside of the tube is cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube is inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation is checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding is to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: Oro-esophageal Feeding
Dietary Supplement: Nasogastric Feeding — Within 4 hours after admission, the placement of the feeding tube is conducted by professional medical staffs and after intubation, the tube is secured to the patient cheek. The feeding is conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements.
  Arms: Nasogastric Feeding

SUMMARY:
This is an open-label randomized controlled trial. The participants are ischemic stroke patients requiring enteral nutrition. The study is conducted in the Department of Rehabilitation Medicine and Department of Neurology.

The purpose of this study is to explore the effects of Intermittent Oro-esophageal Tube Feeding versus Nasogastric Tube Feeding on participants' swallowing function and airway protection.

Specifically, the study aims to answer the following two key questions:

Is there any difference between the two feeding methods in terms of their effects on swallowing function? Are the safety profiles of the two feeding methods consistent? Compared to Nasogastric Tube Feeding, can the Intermittent Oro-esophageal Tube Feeding better improve the nutritional status, extubation of tracheostomy tube, pulmonary infection, neurological deficit of Patients with Intracerebral Hemorrhage Compared to Nasogastric Tube Feeding, is the Intermittent Oro-esophageal Tube Feeding safer.

Participants will be divided into two groups randomly, with different nutritional support respectively.

DETAILED DESCRIPTION:
This is a two-arm open-label randomized controlled trial. The participants are dysphagic ischemic stroke patients requiring enteral nutrition. The study is conducted in the Department of Rehabilitation Medicine and Department of Neurology.

The purpose of this study is to explore the effects of Intermittent Oro-esophageal Tube Feeding versus Nasogastric Tube Feeding on participants' swallowing function and airway protection.

Specifically, the study aims to answer the following two key questions:

Is there any difference between the two feeding methods in terms of their effects on swallowing function? Are the safety profiles of the two feeding methods consistent? Compared to Nasogastric Tube Feeding, can the Intermittent Oro-esophageal Tube Feeding better improve the nutritional status, extubation of tracheostomy tube, pulmonary infection, neurological deficit of Patients with Intracerebral Hemorrhage Compared to Nasogastric Tube Feeding, is the Intermittent Oro-esophageal Tube Feeding safer.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for ischemic stroke.
* Patients who need enteral feeding.
* Dysphagia confirmed by Videofluoroscopic Swallowing Study.
* Clear consciousness.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | Day 0 and day 15
  The Penetration-Aspiration Scale is for assessing airway protection. It has 8 grades, grouped into 3 categories: no penetration/aspiration, penetration, aspiration. Lower grades = better function: Grade 1 is optimal (no airway entry); Grade 8 is most severe (food enters airway below vocal cords with no clearing effort).
Dysphagia Outcome and Severity Scale | Day 0 and day 15
  The Dysphagia Outcome and Severity Scale is a key tool for grading the severity of swallowing disorders and evaluating functional outcomes in patients. It has 7 grades, ranging from severe swallowing impairment to normal swallowing function. Higher grades = better function: Grade 1 means no safe oral intake at all; Grade 7 represents normal swallowing with no restrictions or compensatory strategies.

SECONDARY OUTCOMES:
Functional Oral Intake Scale | Day 0 and day 15
  The Functional Oral Intake Scale is a key tool for grading oral intake ability in patients with swallowing disorders. It has 7 grades, ranging from complete non-oral intake to full oral intake with no restrictions. Higher grades = better function: Grade 1 means total reliance on tube feeding; Grade 7 represents unrestricted oral intake of all consistencies.

OTHER OUTCOMES:
Adverse Events | From day 0 to the end of the study (day 15)
  Both patients and staff are permitted to report any adverse events, which will be documented, categorized and statistically analyzed by the researchers.